CLINICAL TRIAL: NCT01888679
Title: Influence of Head Positioning on the Movement of the Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Patrick Schoettker,MD PD, MD, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 229/12
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: Airway; Endotracheal intubation; selective intubation
MeSH Terms: interventions — Head Movements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- head movement (Experimental): head movement in extension, flexion, right and left rotation
  Interventions: Procedure: Head movement

INTERVENTIONS:
Procedure: Head movement — Head movement in extension, flexion, right and left rotation

SUMMARY:
The purpose of this study is to evaluate and measure the movement of the endotracheal tube depending on the type and the amount of movement of the head of the patient intubated using a flexible fiberoptic.

DETAILED DESCRIPTION:
We performed a maximal head-neck movement trial on 50 adult patients, American Society of Anaesthesiologists 1 or 2. Patients with body mass index N35 kg · m-2, height b150 cm, airway malformations, pulmonary diseases, difficulties in neck flexion or extension, previous ENT surgery or radiotherapy, gastroesophageal reflux, or dental instability were excluded from the study.

We measured the change in distance between the ETT tip and the carina, using a fiberscope through the ETT.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years
* ASA 1-2
* Elective surgery

Exclusion Criteria:

* Pathological changes of the trachea.
* Less than BMI 35 kg/m2.
* Patients with rheumatoid arthritis or other limitation to cervical mobility.
* Emergency surgery.
* Individuals measuring less than 150 cm.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Displacement of the endotracheal tube. | 24 hours
  Tube movement related to movement of the head

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Tailleur R, Bathory I, Dolci M, Frascarolo P, Kern C, Schoettker P. Endotracheal tube displacement during head and neck movements. Observational clinical trial. J Clin Anesth. 2016 Aug;32:54-8. doi: 10.1016/j.jclinane.2015.12.043. Epub 2016 Mar 22. PMID 27290945